CLINICAL TRIAL: NCT00485329
Title: A Phase I/II Randomized, Double Blind, Placebo-Controlled Dose- Escalating Study, to Assess The Safety and Efficacy of Enzystream™ Debriding Solution (Papain) Applied by Dermastream™ Device for the Treatment of Lower Extremity Chronic Venous Ulcers
Brief Title: Assessment of the Safety and Efficacy of DERMASTREAM™ - ENZYSTREAM™ System for the Treatment of Chronic Venous Ulcers
Acronym: ENZ-DER-002-IL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EnzySurge (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENZ-DER-002-IL
Record Dates: First submitted 2007-06-10; First posted 2007-06-12 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Lower Extremity Chronic Venous Ulcers
Keywords: Chronic Wounds, Venous Ulcers, Papain, Debridement, Continuous streaming; DermaStream-EnzyStream
MeSH Terms: conditions — Varicose Ulcer | interventions — Papain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose papain (Experimental): Ratio of drug to placebo treated patients will be 4:1
  Interventions: Other: Papain
- Medium dose papain (Experimental): Ratio of drug to placebo treated patients will be 4:1
  Interventions: Other: Papain
- High dose papain (Experimental): Ratio of drug to placebo treated patients will be 4:1
  Interventions: Other: Papain

INTERVENTIONS:
Other: Papain — 15,000 USP U/ml
  Arms: Low dose papain
Other: Papain — 30,000 USP U/ml
  Arms: Medium dose papain
Other: Papain — 60,000 USP U/ml
  Arms: High dose papain

SUMMARY:
The study objectives are to evaluate DermastreamTM - EnzystreamTM system safety, tolerability and efficacy, as a potent method for debridement of nonhealing lower extremity chronic venous ulcers patients.

DETAILED DESCRIPTION:
This is a phase I/II prospective, randomized, double blind, placebo controlled, dose escalating, three patient-group study, to evaluate the safety and efficacy of DermaStream™ - EnzyStream™ System in non-healing lower extremity chronic venous ulcers patients. The DermaStream™ - EnzyStream™ System will be evaluated during continues streaming of 3 different doses of EnzystreamTM (papain based) solution given in an escalating order (15,000, 30,000 and 60,000 papain USP units/ml) up to 5 consecutive treatment days. Each treatment session lasts for 6 hours. This study is a Multi center trial. It is anticipated that three (3) sites will enroll subjects into this study. Overall, forty eight (48) patients will be recruited, and randomly allocated to placebo or EnzyStream™ treatment in each study dose group prior to EnzyStream™ administration. The ratio of drug to placebo treated patients will be 4;1, namely 12 patients will be administered with EnzyStream™ solution and 4 patients will be placebo treated in each of the three respective EnzyStream™ dose groups. Treatment will start with the lowest dose (15,000 papain USP units/ml) administered over a 6 hour period followed with saline wash for an additional half an hour. The treatment dose will be increased to the next highest dose, for the next patients group only following safety analysis, and the procedure will be repeated.

The treatment period will be followed by a 3 month follow up period. During the follow up period patients will be observed for every 2 weeks during the first month and once a month (every 20 days) during the 2 additional months (allowing a time window of ± 3 days).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a venous leg ulcer
2. Participants, either men or women are between 18 and 85 years of age.
3. Clinical presentation of venous insufficiency demonstrated by Doppler
4. Ankle-Brachial Index > 0.7 by Doppler
5. Good palpable pulses in the Posterior Tibial and the Dorsalis Pedis arteries.
6. Wound present for at least 6 weeks prior to enrolment.
7. Wound length is in the range of: 1.5 - 7 centimeters.
8. The necrotic tissue area is at least 20% of wound area. (by clinical evaluation, i.e., inspection).
9. Wound San Antonio classification: Grade 1 or 2, Stage A or B.
10. Wound location: foot or calf, at a location where the device can be attached properly.
11. Participant understands the nature of the procedure and provides written informed consent prior to any study procedure.
12. Women of child bearing potential must use adequate birth-control precautions.

Exclusion Criteria:

1. Documented sensitivity to Papain, by medical history records.
2. Patients in need of surgical debridement.
3. Patients with general skin disorders (Psoriasis, Peniculitis ect) that might deteriorate as a result of local trauma.
4. Patients with skin disorders unrelated to the ulcer that are presented adjacent to the wound.
5. Pain sensation is completely absent (wound area is anesthetic).
6. Patients with renal failure. (Cr > 2 mg/dl).
7. Patients with impaired hepatic function (ALT, AST or GGT 2-fold higher than normal upper limit value).
8. Patients having Hypoalbuminemia: (Albumin < 2gr/dl ).
9. Patients with general Immunological disorders that might deteriorate as a result of local trauma.
10. Right-side congestive heart failure (CHF) with edema of legs: (NYHA class 2 or higher see APPENDIX 5).
11. Participation in another clinical trial within 1 month prior to start of this study.
12. Subject unwilling or unable to comply with the requirements of the protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To demonstrate Dermastream-Enzystream safety | Up to 88 days
  Skin irritation score
To demonstrate Dermastream-Enzystream safety | Up to 88 days
  Severity and incidence of adverse events
To demonstrate Dermastream-Enzystream safety | 5 days
  No deterioration in clinical laboratory parameters

SECONDARY OUTCOMES:
•Assessment of changes in wound debridement status during treatment period | Days 1-5
  Change in non viable tissue area
Assessment of wound closure | Up to 88 days
  Reduction of nonviable tissue area
Assessment of wound closure | Up to 88 days
  Increase of granulation tissue area
Assessment of wound closure | Up to 88 days
  Time (in days) for wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Arie Bass, Prof., Principal Investigator — Assaf Harofe Medical Center; Sami Nitezki, Dr., Principal Investigator — Rambam Health Care Campus
Locations (3):
- Israel (3):
  - Assaf Harofe Medical Center, Zriffin, Israel
  - Hillel Yafe Medical Center, Hadera
  - Rambam Medical Center, Haifa